CLINICAL TRIAL: NCT02312076
Title: Gonadotropin Releasing Hormone Agonist for Luteal Phase Support in Long Gonadotropin Releasing Hormone Agonist Protocol Cycles
Brief Title: GnRHa for Luteal Phase Support in Long GnRHa Protocol Cycles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSA3
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Infertility
Keywords: Luteal phase support, ICSI, GnRHa
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GnRHa group (Active Comparator): Luteal phase SC administration of a single dose (0.2 mg) of GnRHa (Triptorelin)
  Interventions: Drug: Triptorelin
- Control group (No Intervention): No GnRHa administration in luteal phase

INTERVENTIONS:
Drug: Triptorelin — Luteal phase support will be continued by the same regimen started on the day of oocytes retrieval until 2 weeks after embryo transfer (ET) with subcutaneous administration of a single dose (0.2 mg) of GnRHa (Triptorelin) 6 days after oocyte retrieval
  Other Names: Decapeptyl
  Arms: GnRHa group

SUMMARY:
Evaluation of the effect of adding a single dose of gonadotropin releasing hormone agonist (GnRHa) as a luteal phase support on the outcomes of intracytoplasmic sperm injection (ICSI) following long GnRHa protocol

DETAILED DESCRIPTION:
Endometrial preparation for embryo transfer (ET) will be started after oocyte retrieval by giving 800 mg/day natural progesterone vaginal supplement + 4 mg/day estradiol oral supplement. The patients will be randomly divided into 2 groups for luteal phase support: (i) Group A (GnRHa group) in which the luteal phase support will be continued by the same regimen started on the day of oocytes retrieval until 2 weeks after embryo transfer (ET) with subcutaneous administration of a single dose (0.2 mg) of GnRHa (Triptorelin) 6 days after oocyte retrieval, and (ii) Group B (control group) in which the luteal phase support will be continued only by the same regimen started on the day of oocytes retrieval until 2 weeks after ET

ELIGIBILITY:
Inclusion Criteria:

* Women subjected to ICSI through controlled ovarian hyperstimulation (COH) with pituitary downregulation by GnRHa.

Exclusion Criteria:

* Moderate or severe endometriosis.
* Hydrosalpinx.
* Uterine abnormalities.
* Myoma.
* Previous uterine surgery.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 4-6 weeks after the ET) divided by the number of ET procedures

SECONDARY OUTCOMES:
Implantation rate | 6 weeks after embryo transfer
  Number of gestational sacs on TVS scan at 4-6 weeks after ET divided by the number of transferred embryos
Miscarriage rate | 12 weeks gestational age
  Number of first trimester miscarriages (before 12 weeks gestational age) divided by the number of clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Abdelhafez, Dr, Principal Investigator — Mansoura University
Locations (2):
- Egypt (2):
  - Fertility Care Unit (FCU) in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private fertility care centers, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: No